CLINICAL TRIAL: NCT06814743
Title: Analysis, Awareness and Tele-rehabilitation of Urinary Incontinence and Other Pelvic Floor Dysfunctions in Female Athletes
Brief Title: A Mobile Application for Female Athletes With Pelvic Floor Dysfunctions (ACTITUD2.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Ministerio de Ciencia, Innovación y Universidades, Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 124CER19_2.0
Record Dates: First submitted 2025-01-21; First posted 2025-02-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Floor Disorders
Keywords: Female; Athletes; e-Health; Exercises
MeSH Terms: conditions — Pelvic Floor Disorders; Motor Activity | interventions — Health Personnel

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The design of this study does not allow to mask participants or care providers. Investigators and outcomes assessors will not know which group athletes belong to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 2: Exercises with biofeedback guidance (Experimental): All participants will use a mobile application with access to information about pelvic floor and communication with healthcare team, and a exercise program for pelvic floor, while using an intravaginal biofeedback device.
  Interventions: Behavioral: Pelvic floor exercises program guided with an intravaginal biofeedback device; Behavioral: Pelvic floor exercises program; Behavioral: Information about pelvic floor and communication with health professionals
- Experimental group 1: Exercises (Active Comparator): All participants will use a mobile application with access to information about pelvic floor and communication with healthcare team, and a exercise program for pelvic floor.
  Interventions: Behavioral: Pelvic floor exercises program; Behavioral: Information about pelvic floor and communication with health professionals
- Control group: No exercises (Active Comparator): All participants will use a mobile application with access to information about pelvic floor and communication with healthcare team.
  Interventions: Behavioral: Information about pelvic floor and communication with health professionals

INTERVENTIONS:
Behavioral: Pelvic floor exercises program guided with an intravaginal biofeedback device — Use of the mobile application to perform a exercise program for pelvic floor musculature, while using an intracavitary biofeedback device that will inform about vaginal pressure. Behavioral: mobile application with access to information about pelvic floor and direct communication with healthcare team.
  Other Names: Information about pelvic floor and communication with health professionals
  Arms: Experimental group 2: Exercises with biofeedback guidance
Behavioral: Pelvic floor exercises program — Use of the mobile application to perform a exercise program for pelvic floor musculature.
  Behavioral: Information about pelvic floor and communication with health professionals Use of the mobile application with access to information about pelvic floor and direct communication with healthcare team.
  Other Names: Information about pelvic floor and communication with health professionals
  Arms: Experimental group 1: Exercises; Experimental group 2: Exercises with biofeedback guidance
Behavioral: Information about pelvic floor and communication with health professionals — Use of the mobile application with access to information about pelvic floor and direct communication with healthcare team.

SUMMARY:
Pelvic floor dysfunctions (PFD) are especially prevalent among females. As conservative management, strengthening pelvic floor (PF) musculature under health supervision, regard an important research line. However, embarrassment of female athletes limits healthcare demands. New technologies could facilitate an autonomous but supervised tele-rehabilitation programs.

This study will evaluate the effects of a 12-weeks program with exercises focused on PF awareness and strengthening by using a mobile application supervised by physiotherapists, with or without intracavitary biofeedback, on the PF anatomical and functional characteristics, symptomatology and sports performance of female athletes with PFD.

To this end, 105 female athletes with self-reported PFD who train and compete in sport in Spain will be recruited and randomly distributed in three groups of the experimental study. During 12 weeks, all participants will use the mobile application (named ACTITUD): the control group (CG) will have access to information about PF and direct communication with healthcare team; experimental group 1 (EG1) will have access to the same information and communication, and will perform a the exercise program for PF; the experimental group 2 (EG2) will be similar to EG1, but they will use an intravaginal biofeedback device during exercises to receive information about their intra-vaginal pressure.

Before and after these 12 weeks, anatomical and functional PF characteristics, PF symptoms and sports performance of all participants will be evaluated. As additional outcome, the compliance of the athletes from experimental groups to complete the training program will be registered (in %).

DETAILED DESCRIPTION:
Female athletes from EG1 and EG2 will complete the exercise program for PF three times per week, during 12 weeks. Each session will last about 20 minutes and exercises will be modified every two weeks to meet the principle of training progression and avoid athletes become bored.

ELIGIBILITY:
Inclusion Criteria:

* To train and compete in any sport.
* To have a self-reported pelvic floor disorder (urinary incontinence, anorectal incontinence, sexual dysfunction or chronic pelvic pain).

Exclusion Criteria:

* To have recurrent infections of urinary tract during the last three months.
* To be receiving physiotherapy treatment due to any pelvic floor disorder at the moment of the start of the study.
* To have been pregnant during the year prior to the start of the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Functional characteristics of pelvic floor musculature | 12 weeks
  Change in the pelvic floor strength according to the modified grading Oxford Scale (graded from 0 - minimal strength- to 5 points - maximal strength) after the intervention period and compared to the athletes from the rest of groups. To assess it, the evaluator will insert the first two phalanges of the second and third fingers smeared in lubricant gel with a gloved hand into the anterior third of the vaginal opening and will request a maximal voluntary contraction (MVC) by giving the command "contract the anus, do as if you wanted to hold a strong desire to void".
Functional characteristics of pelvic floor musculature with manometry I | 12 weeks
  Change in the maximal voluntary contraction (MVC) according to the values of pressure collected by a manometer (in cmH20) after the intervention period and compared to the athletes from the rest of groups. To assess it, participants will perform a maximal contraction of pelvic floor musculature during 3 seconds (two trials with 30 seconds apart). The best trial (the highest pressure) will be collected.
Functional characteristics of pelvic floor musculature with manometry II | 12 weeks
  Change in the vaginal pressure at rest (in cmH20) after the intervention period and compared to the athletes from the rest of groups. To assess it, the probe of the manometer will be covered with a lubricated condom and placed about 3.5 cm proximal to the vaginal introitus, without pain or discomfort. The air in the probe will be emptied before being inserted into the vagina introitus and vaginal pressure at rest will be registered.
Functional characteristics of pelvic floor musculature with manometry III | 12 weeks
  Change in the proprioceptive error during a force sense test (Proprioception) according to the values of pressure collected by a manometer (in cmH20) after the intervention period and compared to the athletes from the rest of groups. To assess it, participants will perform a contraction of pelvic floor musculature at 50% of maximal voluntary contraction (MVC) (TARGET) during 3 seconds (two trials with 10 seconds apart). The difference between the average of the two trials and the target value will be the proprioceptive error (in %).
Anatomical characteristics of pelvic floor structures with ultrasound I | 12 weeks
  Change in the levator hiatus length (in mm) after the intervention period and compared to the athletes from the rest of groups. This variable will be assessed by using transperineal approach with transducer in longitudinal orientation, at three different functional situations: at rest, while participants perform a maximal voluntary contraction (MVC) of the pelvic floor musculature, and also at straining.
Anatomical characteristics of pelvic floor structures with ultrasound II | 12 weeks
  Change in the anorectal angle (in degrees) and pubourethral angle (in degrees) after the intervention period and compared to the athletes from the rest of groups. These variables will be assessed by using transperineal approach with transducer in longitudinal orientation, at three different functional situations: at rest, while participants perform a maximal voluntary contraction (MVC) of the pelvic floor musculature, and also at straining.
Anatomical characteristics of pelvic floor structures with ultrasound III | 12 weeks
  Change in the symmetry of the bladder base (in mm) at rest and bladder base displacement (in mm) while participants perform a maximal voluntary contraction (MVC) of the pelvic floor musculature and also during straining, after the intervention period and compared to the athletes from the rest of groups. These variables will be assessed by using a transabdominal approach with transducer, in transverse orientation.
Sports performance through maximal vertical jump I | 12 weeks
  Change in the maximal height that athletes reach with a vertical jump (in meters) after the intervention period and compared to the athletes from the rest of groups. To assess it, participants will perform a maximal countermovement jump (three trials with 60 seconds apart). It will be collected the best of the three trials.
Sports performance through maximal vertical jump II | 12 weeks
  Change in the maximal ground reaction forces during a vertical jump (in Newton) after the intervention period and compared to the athletes from the rest of groups. To assess it, participants will perform a maximal countermovement jump (three trials with 60 seconds apart). It will be collected the best of the three trials.
Occurrence of urinary incontinence symptomatology | 12 weeks
  Change in self-reported pelvic floor symptoms regarding urinary incontinence, assessed through the International Consultation on Incontinence Questionnaire - Short form (ICIQ-SF) after the intervention period and compared to the athletes from the rest of groups. To this end, athletes will reply the proposed tool consisting of 3 questions, with a total score of 21 points. Scoring 0 points will mean that athletes do not have urinary incontinence; score between 1 and 21 will mean a progressively more severe urinary incontinence.
Sexual dysfunction symptomatology | 12 weeks
  Change in self-reported sexual dysfunction symptoms (orgasm and pain domains of the Female Sexual Function Index - FSFI), after the intervention period and compared to the athletes from the rest of groups. The score of each domain is rated from 1 (the worst sexual function) to 15 points (the best sexual function)
Occurrence of ano-rectal incontinence | 12 weeks
  Change in self-reported pelvic floor symptoms regarding ano-rectal incontinence, assessed through the Wexner Scale, after the intervention period and compared to the athletes from the rest of groups. To this end, athletes will reply the proposed tool consisting of 5 questions ranging from 0 (never incontinent) to 4 (always incontinent). A score of 0 points will mean that athletes do not have ano-rectal incontinence. Results in the score from 1 to 20 will mean ano-rectal incontinence progressively more severe.
Level of quality of life | 12 weeks
  It will be explore the change in quality of life due to the pelvic floor disorders symptoms (according to a scale from 0, no affection, to 10, maximal affection) after the intervention period and compared to the athletes from the rest of groups.

SECONDARY OUTCOMES:
Compliance to the proposed pelvic floor exercise program | 12 weeks
  Percentage of exercises program sessions that athletes from experimental groups 1 and 2 completed during the 12 weeks of intervention, according to the number of proposed sessions (three times per week).

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Romero-Franco, Principal Investigator — University of the Balearic Islands; Natalia Romero-Franco, PhD, Principal Investigator — University of the Balearic Islands
Locations (1):
- Palma de Mallorca, Palma, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No